CLINICAL TRIAL: NCT04194255
Title: The Effect of Single Dose Oral Galacto-oligosaccharides, Fructo-oligosaccharides and Acacia Gum on Iron Absorption From Single 100 mg Oral Iron Doses Given as Ferrous Fumarate in Women Living in Switzerland
Brief Title: The Effect of Different Prebiotics on Iron Absorption From High Dose Iron Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: HIGH
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Iron-deficiency
Keywords: iron-deficiency; Prebiotics; galacto-oligosaccharides; fructo-oligosaccharides; acacia gum
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferrous fumarate; Gum Arabic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ferrous fumarate (Experimental): labelled iron as ferrous fumarate
  Interventions: Dietary Supplement: ferrous fumarate
- ferrous fumarate + 15 g GOS (Experimental): labelled iron as ferrous fumarate + prebiotics in the form of 15 g GOS
  Interventions: Dietary Supplement: ferrous fumarate + 15 g GOS
- ferrous fumarate + 15 g FOS (Experimental): labelled iron as ferrous fumarate + prebiotics in the form of 15 g FOS
  Interventions: Dietary Supplement: ferrous fumarate + 15 g FOS
- ferrous fumarate + 15 g acacia gum (Experimental): labelled iron as ferrous fumarate + prebiotics in the form of 15 g acacia gum
  Interventions: Dietary Supplement: labelled iron as ferrous fumarate + 15 g acacia gum

INTERVENTIONS:
Dietary Supplement: ferrous fumarate — iron (100 mg) supplement in form of ferrous fumarate
  Arms: ferrous fumarate
Dietary Supplement: ferrous fumarate + 15 g GOS — iron (100 mg) supplement in form of ferrous fumarate with addition of prebiotics (15 g GOS)
  Arms: ferrous fumarate + 15 g GOS
Dietary Supplement: ferrous fumarate + 15 g FOS — iron (100 mg) supplement in form of ferrous fumarate with addition of prebiotics (15 g FOS)
  Arms: ferrous fumarate + 15 g FOS
Dietary Supplement: labelled iron as ferrous fumarate + 15 g acacia gum — iron (100 mg) supplement in form of ferrous fumarate with addition of prebiotics (15 g acacia gum)
  Arms: ferrous fumarate + 15 g acacia gum

SUMMARY:
Iron deficiency (ID) remains the most common global nutrient deficiency, with young women at high risk. Iron supplements are first line treatment for ID but absorption is often low. Dietary components that could increase iron absorption would be valuable.

Prebiotics are among the potential enhancers of non-heme iron absorption. Galacto-oligosaccharides (GOS), fructo-oligosaccharides and acacia gum are safe and widely-used prebiotics.

To our knowledge, no studies have assessed the effect of acacia gum on iron absorption in human or animal models. Evidence exists about the enhancement of iron absorption when given in combination with FOS in rats. However, an iron stable isotope study in infants reported that 7.5 g of GOS improved iron absorption from 5 mg iron from a mixture of ferrous fumarate and sodium iron EDTA. In a recent iron absorption study in adult women with low iron stores in our lab we found that 15 g of GOS given with FeFum (14 mg of elemental iron) acutely increased iron absorption when given with water (+61%) and a meal (+28%).

For prevention of anemia among non-pregnant women, the WHO recommends intermittent (once, twice or three times a week) oral iron supplementation with 60 mg of elemental iron. This has been shown to be effective, safe and acceptable for improving hemoglobin concentrations in women and lowering their risk of anemia. If GOS improves iron absorption from a higher dose of iron, and if FOS and acacia gum might also enhance iron absorption from FeFum is unclear. With this study we therefore aim to investigate if consumption of a single oral dose of 15 g GOS, FOS or acacia gum increase iron absorption from single 100 mg oral iron doses, a common amount found in supplements on the market for treatment of iron deficiency, given as ferrous fumarate in otherwise healthy iron depleted women.

DETAILED DESCRIPTION:
Prebiotics are defined as "microbial food supplements that beneficially affect the host by selectively stimulating the growth and/or activity of one or a limited number of bacterial species already resident in the colon". Moreover, prebiotics are potential enhancers of iron absorption, via several mechanisms: a) increasing gastric residence time allowing for greater iron dissolution; b) stimulating enterocyte gene expression of proteins involved in iron absorption; c) stimulating enterocyte proliferation providing a greater surface for iron absorption; and d) stimulating SCFA production by gut commensal bacteria, decreasing distal gut luminal pH and increasing iron dissolution.

Galacto-oligosaccharides (GOS), a safe and widely-used prebiotic, are a mixture of glucose- and galactose-based di- and oligosaccharides of varying structure and may be more selectively utilized by Bifidobacterium spp. than other prebiotics. Fructo-oligosaccharides (FOS) are composed by 4 to 9 units of fructose alone or in combination with one unit of glucose. FOS are widely used as food ingredients/nutritional supplements due to their bifidogenic properties. Acacia gum is composed by highly branched galactan polymers with galactose and/or arabinose side chains, possibly terminated by rhamnose or glucuronic acid residues. Both in-vitro and in-vivo studies have shown that acacia gum supports bifidobacterial growth and short-chain fatty acids (SCFA) production in the large intestine.

GOS and FOS have received GRAS status in the USA. Acacia gum is extensively used in the food industry for various functions (emulsification, encapsulation, stabilization, etc.). It is affirmed as "GRAS" for use in various food items. Acacia gum in human subjects is well tolerated up to 50 g/day. The European Food Safety Authority stated that there is no safety concern for the use of Acacia Gum as a food supplement.

To our knowledge, no studies have assessed the effect of acacia gum on iron absorption in human or animal models. Evidence exists about the enhancement of iron absorption when given in combination with FOS in rats. In humans, studies so far have failed in showing an effect of FOS on iron absorption. However, an iron stable isotope study in infants reported that 7.5 g of GOS improved iron absorption from 5 mg iron from a mixture of ferrous fumarate and sodium iron EDTA. Moreover, in a recent iron absorption study in adult women with low iron stores in our lab we found that 15 g of GOS given with FeFum (14 mg of elemental iron) acutely increased iron absorption when given with water (+61%) and a meal (+28%). In another study in our lab (unpublished data) we found that 7 g of GOS given with FeFum (14 mg of elemental iron) acutely increased iron absorption when given with water (+26%), in iron depleted women. These effects were found to be iron compound specific and could not be shown for ferrous sulfate, the iron compound used in the existing human studies with FOS.

For prevention of anemia among non-pregnant women, the WHO recommends intermittent (once, twice or three times a week) oral iron supplementation with 60 mg of elemental iron. This has been shown to be effective, safe and acceptable for improving hemoglobin concentrations in women and lowering their risk of anemia.

If GOS improves iron absorption from a higher dose of iron, and if FOS and acacia gum might also enhance iron absorption from FeFum is unclear. With this study we therefore aim to investigate if consumption of a single oral dose of 15 g GOS, FOS or acacia gum increase iron absorption from single 100 mg oral iron doses, a common amount found in supplements on the market for treatment of iron deficiency, given as ferrous fumarate in otherwise healthy iron depleted women.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 45 years old
* SF concentrations ≤ 25 µg/L
* Normal body Mass Index (18.5-24.9 kg/m2)
* Body weight <70 kg
* Signed informed consent

Exclusion Criteria:

* Anaemia (Hb < 11,7g/dL)
* Any metabolic, gastrointestinal, kidney or chronic disease such as diabetes, renal failure, hepatic dysfunction, hepatitis, hypertension, cancer or cardiovascular diseases (according to the participants own statement)
* Continuous/long-term use of medication during the whole study (except for contraceptives),
* Consumption of mineral and vitamin supplements within 2 weeks prior to 1st supplement administration, including pre- and/or probiotic supplements (excluding foods and beverages with life cultures such as yoghurt, raw milk cheese and kombucha)
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 4 months
* Known difficulties with blood sampling
* Use of antibiotics over the past month
* Known hypersensitivity to iron supplements in the given amount, GOS, or lactose
* Women who are pregnant or breast feeding
* Women who intend to become pregnant during the course of the study
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases
* Known or suspected non-compliance, drug or alcohol (more than 2 drinks/day) abuse
* Smokers (> 1 cigarette per week)
* Inability to follow the procedures of the study, e.g. due to language problems, self-reported psychological disorders, etc. of the participant
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female participants are being studied
Enrollment: 30 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
fractional iron absorption | 43 days
  Fractional iron absorption will be calculated based on the shift of the iron isotope ratios in the collected blood samples after the administration of several isotopically labelled iron supplements.Fractional iron absorption will be measured as erythrocyte incorporation of the naturally occurring iron forms with different masses used to label the iron supplements.

SECONDARY OUTCOMES:
Hemoglobin (Hb) | Baseline, 43 days
Serum ferritin | Baseline, 43 days
soluble transferrin receptor | Baseline, 43 days
serum iron | Baseline, 43 days
alpha-1-acid glycoprotein (AGP) | Baseline, 43 days
C-reactive protein (CRP) | Baseline, 43 days
Retinol binding protein (RBP) | Baseline, 43 days

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Herter-Aeberli, PhD, Study Director — Laboratory of Human Nutrition ETH Zürich
Locations (1):
- Human Nutrition Laboratory, ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giorgetti A, Husmann FMD, Zeder C, Herter-Aeberli I, Zimmermann MB. Prebiotic Galacto-Oligosaccharides and Fructo-Oligosaccharides, but Not Acacia Gum, Increase Iron Absorption from a Single High-Dose Ferrous Fumarate Supplement in Iron-Depleted Women. J Nutr. 2022 Apr 1;152(4):1015-1021. doi: 10.1093/jn/nxac003. PMID 35015879